CLINICAL TRIAL: NCT04435509
Title: Randomized, Double Blind, Placebo Controlled Prospective Study, to Evaluate the Effect of Greek Mountain Tea Patiens With Mild Cognitive Impairment
Brief Title: Management of Mild Cognitive Impairment Patients With Greek Mountain Tea - TEAMENTIA
Acronym: TEAMENTIA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Magda Tsolaki, MD, PhD, Professor, President of Greek Alzheimer's Association and Related Disorders, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 31c/17-05-17
Record Dates: First submitted 2019-10-08; First posted 2020-06-17 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment,; Intervention; Greek Mountain Tea
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Diet, Mediterranean

STUDY DESIGN:
Intervention Model Description: Single (Participant)
Who Masked: Participant
Masking Description: Single (Participant)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Greek Mountain Tea (Experimental): 50 patients Greek Mountain Tea 50 grams one per 30 days. Dietary Supplement: Greek Mountain Tea dietary intake of the content of 12 grams Intervention:Greek Mountain Tea in a plastic bag.
  Interventions: Dietary Supplement: 1000+ Greek Mountain Tea
- Mediterranean Diet (Placebo Comparator): 50 patients same dietary habits and a Mediterranean dietary protocol Intervention: Mediterranean diet.
  Interventions: Other: Mediterranean Diet

INTERVENTIONS:
Dietary Supplement: 1000+ Greek Mountain Tea — Dietary Supplement: Greek Mountain Tea dietary intake of the content of 12 grams (4 grams 3 times per day ) 50 grams per month
  Arms: Greek Mountain Tea
Other: Mediterranean Diet — a Mediterranean dietary protocol
  Arms: Mediterranean Diet

SUMMARY:
There is accumulating evidence suggesting that Greek Mountain Tea may have a positive impact on conditions involving cognitive deficits, such as Mild Cognitive Impairment (MCI) and AD. More specifically, greek mountain olympos tee is rich in essential oils, flavonoids, diterpenes and phenylpropanes, which are primarily responsible for its pharmacological properties. Its confirmed antioxidant properties are what make mountain tea promising against Alzheimer's disease and other neurodegenerative diseases. It has also been proven to possess cholinergic and cognitive enhancing capabilities. Greek Mountain Tea is deeper studied and it shows promising results in neuroprotection against AD through various suggested mechanisms, such as the enhancement of amyloid-beta clearance in the brain and the inhibition of neurofibrillary tangles formation. The aim of the study is to evaluate the beneficial effect of Greek Mountain Tea in patients diagnosed with mild cognitive impairment MCI.

Study Type: Interventional Study Design: Allocation: Randomized Intervention Model: Parallel Assignment Masking: Double Blind (Subject, Investigator) Primary Purpose: Prevention

DETAILED DESCRIPTION:
OBJECTIVES OF THE TRIAL

The objectives of this study are:

To investigate the efficacy of Greek Mountain Tea as a disease course modifying treatment for MCI in a phase III double-blind placebo-controlled study.

To investigate the effects in objective measurements in patients with MCI.

STUDY DESIGN This is a Greek, randomised, double-blind, placebo-controlled study group of compared Greek Mountain Tea placebo. Qualifying patients will be randomly assigned to receive 12 grams of Greek Mountain Tea or mediterranean dietary protocol on a daily basis for 24 months. Patients undergo assessments at baseline,12 and 24 months +/- 7 days after beginning of the treatment.

Duration The total study duration will be 36 months. Patients will receive study medication for 24 months.The recruitment will be about 6 months and the statistics and the preparation of the paper other 6 months. Number of Subjects One hundred fifty (100) subjects total will be enrolled. ; Fifty (50) in the experimental group (Greek Mountain Tea); and Fifty (50) in control Group 2(same dietary habits mediterranean dietary protocol).

Patient Eligibility Screening Form (ESF)

An eligibility form documenting the patient's fulfilment of the entry criteria will be completed by the assessor. The following information will be included in the

ESF:

Patient identification: Initials (First initial of first name and First initial of surname), date of birth and Patient Identification Number.

Eligibility Screening; Checklist of inclusion and exclusion criteria Eligibility Statement; for patients found to be ineligible, the reason for ineligibility must be stated Written informed consent will be obtained from the subject . The informed consent form must be co-signed by the physician. The nature of the study and the potential risks associated with the trial will be explained to all subject candidates and their responsible informants.

Signature and date: the ESF may be completed by an assessor but it is required that the principal investigator/study clinician sign and date the ESF to verify eligibility of the patient for inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Memory Complaints
* Abnormal memory function documented by scoring 1 SD below the ageadjusted mean on the Logical Memory II subscale, (Delayed Paragraph Recall) from the Wechsler Memory Scale-R.
* MMSE 24-30
* CDR(sum of boxes) >= 0,5
* Diagnosis: Mild Cognitive Impairment (amnestic plus multi-domain)
* Geriatric Depression Scale (GDS) <6
* Hachinski Modified Ischemic scale <= 4
* Stability of Permitted Medications for 4 weeks
* Years of education: >= 5
* Proficient language fluency
* Compliance

  -Exclusion Criteria:
* Antidepressants with anti-cholinergic properties.
* Regular use of narcotic analgesics (>2 doses per week) within 4 weeks of screening.
* Use of neuroleptics with anti-cholinergic properties (e.g., chlorpromazine, thioridazine) within 4 weeks of screening.
* Chronic use of other medications with significant central nervous system anticholinergic activity within 4 weeks of screening (e.g., diphenhydramine).
* Use of Anti-Parkinsonian medications (including Sinemet, amantadine, bromocriptine, pergolide, selegeline) within 4 weeks of screening.
* Participation in any other investigational drug study within 4 weeks of screening (individuals may not participate in any drug study while participating in this protocol).

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-11-17 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2021-05-30 (Estimated)

PRIMARY OUTCOMES:
Neuropsychological Assessment- Measurements to Assess General Cognitive Function | baseline, 12 and 24 months
  Changes in Mini-Mental State Examination (MMSE) score
FUCAS-Measurements to Assess Daily Functionality | baseline, 12 and 24 months
  Changes in Functional cognitive assessment scale (FUCAS) score
Letter & Category Fluency Test- Measurement to Assess Verbal Fluency and Learning | baseline, 12 and 24 months
  Changes in the Letter & Category Fluency Test
CDR- Measurements to Assess General Cognitive Function | baseline, 12 and 24 months
  Changes in Global Clinical Dementia Rating (CDR) score (sum of boxes)
MoCA- Measurements to Assess General Cognitive Function | baseline, 12 and 24 months
  Changes in Montreal Cognitive Assessment (MoCA)
CANTAB- Measurements to Assess General Cognitive Function | baseline, 12 and 24 months
  Changes in Cambridge Neuropsychological Test Automated Battery (CANTAB)
Clock Drawing test- Measurements to Assess General Cognitive Function | baseline, 12 and 24 months
  Changes in the Clock Drawing test
Logical Memory test- Measurements to Assess General Cognitive Function | baseline, 12 and 24 months
  Changes in the Logical Memory test
Digit Span Forward & Backward test- Measurements to Assess General Cognitive Function | baseline, 12 and 24 months
  Changes in the Digit Span Forward & Backward test
WAIS-R Digit Symbol- Measurements to Assess General Cognitive Function | baseline, 12 and 24 months
  Changes in the WAIS-R Digit Symbol Substitution Test
TMT part A and B- Measurements to Assess General Cognitive Function | baseline, 12 and 24 months
  Changes in the Trail Making Test
ADASCog-Measurements to Assess Daily Functionality | baseline, 12 and 24 months
  Changes in Alzheimer's Disease Assessment Scale-Cognitive (ADASCog)
Functional Rating Scale for Dementia-Measurements to Assess Daily Functionality | baseline, 12 and 24 months
  Changes in Functional Rating Scale for Dementia (FRSSD)
Auditory Verbal Learning Test- Measurement to Assess Verbal Fluency and Learning | baseline, 12 and 24 months
  Changes in the Auditory Verbal Learning Test
Boston Naming Test- Measurement to Assess Verbal Fluency and Learning | baseline, 12 and 24 months
  Changes in the Boston Naming Test

SECONDARY OUTCOMES:
NeuroImaging | baseline, 12 and 24 months]
  Changes in brain Magnetic Resonance Imaging (MRI) 1.5 Tesla (brain atrophy)
CSF - beta amyloid | baseline, 12 and 24 months
  Changes in mean values on high sensitivity beta-amyloid 1-42 protein
CSF TAU-protein | baseline, 12 and 24 months
  Changes in mean values on TAU-protein in cerebrospinal fluid
Electroencephalography recording | baseline, 12 and 24 months
  * Changes in Event-Related Potential (ERP) (oddball paradigm, auditory ERPs) Electroencephalography recording
  * Changes in Electroencephalography (EEG), resting state. The device records brain signals through 57 electrodes, 2 reference electrodes attached to the earlobes, and a ground electrode placed at a left anterior position

OTHER OUTCOMES:
Weight in Kilograms | baseline, 12 and 24 months
  Changes in weight
Height in Meters | baseline, 12 and 24 months
  Changes in Height

CONTACTS AND LOCATIONS:
Locations (1):
- Greek Alzheimer's Association and Related Disorders, Thessaloniki, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tsolaki M, Karathanasi E, Lazarou I, Dovas K, Verykouki E, Karacostas A, Georgiadis K, Tsolaki A, Adam K, Kompatsiaris I, Sinakos Z. Efficacy and Safety of Crocus sativus L. in Patients with Mild Cognitive Impairment: One Year Single-Blind Randomized, with Parallel Groups, Clinical Trial. J Alzheimers Dis. 2016 Jul 27;54(1):129-33. doi: 10.3233/JAD-160304. PMID 27472878
- [Result] Tzekaki EE, Tsolaki M, Pantazaki AA, Geromichalos G, Lazarou E, Kozori M, Sinakos Z. Administration of the extra virgin olive oil (EVOO) in mild cognitive impairment (MCI) patients as a therapy for preventing the progress to AD. Hell J Nucl Med. 2019 Sep-Dec;22 Suppl 2:181. PMID 31802059